CLINICAL TRIAL: NCT07192341
Title: Effect of Sacubitril/Valsartan in Patients With Prosthetic Heart Valves With Heart Failure and Reduced Ejection Fraction
Brief Title: Sacubitril/Valsartan in Patients With Prosthetic Heart Valves With Heart Failure and Reduced Ejection Fraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohammed Ali Mohammed Hammad, Lecturer of Cardiology, Faculty of Medicine, Kafr Elsheikh University, Kafr Elsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-728
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Sacubitril/Valsartan; Prosthetic Heart Valve; Heart Failure; Reduced Ejection Fraction
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group S (Experimental): Patients will be treated with conventional anti-heart failure therapy plus sacubitril/valsartan (oral administration of an initial dose of 24/26 mg twice daily, gradually increasing to 97/103 mg, depending on follow-up blood pressure) [Entresto, 100 mg (sacubitril 49 mg/valsartan 51 mg)].
  Interventions: Drug: Sacubitril/Valsartan
- Group C (Active Comparator): Patients will be treated only with conventional anti-heart failure therapy as a control group.
  Interventions: Drug: Conventional anti-heart failure therapy

INTERVENTIONS:
Drug: Sacubitril/Valsartan — Patients will be treated with conventional anti-heart failure therapy plus sacubitril/valsartan (oral administration of an initial dose of 24/26 mg twice daily, gradually increasing to 97/103 mg, depending on follow-up blood pressure) [Entresto, 100 mg (sacubitril 49 mg/valsartan 51 mg)].
  Arms: Group S
Drug: Conventional anti-heart failure therapy — Patients will be treated only with conventional anti-heart failure therapy as a control group.
  Arms: Group C

SUMMARY:
This study aims to evaluate the effect of sacubitril/valsartan in patients with prosthetic heart valves with heart failure with reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
Heart failure (HF) is the end stage of various types of cardiovascular disease. The prevalence of HF continues to rise, and the rates of readmission and mortality also continue to increase significantly.

There are three types of HF, heart failure with preserved ejection fraction (HFpEF), heart failure with mid-range ejection fraction (HFmrEF), and heart failure with reduced ejection fraction (HFrEF).

Sacubitril/valsartan, the first angiotensin receptor-neprilysin inhibitor (ARNI) approved by the FDA for the treatment of HFrEF, demonstrated significant benefits in the PARADIGM-HF trial. PARADIGM-HF trial was a large multicenter, randomized clinical trial comparing sacubitril/ valsartan with enalapril in patients with LVEF < 40%. This trial showed 20% reduction in composite Cardiovascular (CV) death (including sudden cardiac death) and hospitalization for HF patients with S/V.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Both sexes.
* Patients with a history of prosthetic heart valves.
* Patients diagnosed with heart failure with reduced ejection fraction (HFrEF), defined as left ventricular ejection fraction (LVEF) ≤ 40% with New York Heart Association (NYHA) functional class II-IV.

Exclusion Criteria:

* Hemodynamic instability.
* Use of a circulatory auxiliary circulation device.
* Severe hepatic [alanine aminotransferase (ALT) >120 U/L] and renal insufficiency [estimated glomerular filtration rate (eGFR) <30 mL/min].
* Blood pressure <100/60 mmHg.
* Serum potassium >5.3 mmol/L.
* Severe pulmonary hypertension.
* Malignant arrhythmia.
* Malignant tumor.
* Known history of hereditary or primary angioedema.
* Serious adverse drug reactions or serious complications over the course of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-09-27 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Effective rate | 6 months post-procedure
  Effectiveness is defined as an New York Heart Association (NYHA) cardiac function grade improved by 1 grade or more.
  Effective rate= Effectiveness/total quantity*(100%).

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: The data will be available upon a reasonable request from the corresponding author.
Access Criteria: After the end of study for one year.